CLINICAL TRIAL: NCT07208695
Title: Effect of Oral Antiplatelet or Anticoagulant Drugs on Postoperative Bleeding Risk and Venous Closure Rate in Patients With Lower Extremity Varicose Veins After Radiofrequency Ablation
Status: Not yet recruiting | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, chief physician, Chengdu University of Traditional Chinese Medicine
Other Study IDs: ChengduUTCM 276
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Oral Antiplatele; Anticoagulant Drugs; Lower Extremity Varicose Veins; Radiofrequency Ablation
MeSH Terms: interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiplatelet or Anticoagulant Drugs — The goal of this observational study is to assess the effect of postoperative continuous use of standard-dose oral antiplatelet (e.g., aspirin, clopidogrel) or anticoagulant drugs (e.g., warfarin, direct oral anticoagulants) on key postoperative outcomes in patients with primary lower extremity varicose veins who have undergone endovenous radiofrequency ablation (RFA) of the great saphenous vein. Unlike studies focusing on preoperative medication adjustment or single-drug cohorts, this study specifically targets routine postoperative medication use without protocol-mandated dose changes, and distinguishes between two major classes of antithrombotic agents while including a non-user control group. The main questions it aims to answer are: 1) Whether postoperative oral antiplatelet/anticoagulant use correlates with increased 30-day bleeding risk (defined by standardized criteria: minor = localized ecchymosis needing no intervention; major = bleeding requiring transfusion or surgical hemo

SUMMARY:
This observational study aims to assess the effect of oral antiplatelet or anticoagulant drugs on key postoperative outcomes in patients with lower extremity varicose veins who have undergone radiofrequency ablation. Its main objectives are to determine the impact of these medications on postoperative 30-day bleeding risk and postoperative 3-month venous closure rate in this patient population. Researchers will compare three groups-patients receiving oral antiplatelet drugs, those receiving oral anticoagulant drugs, and those not receiving either type of drug-to identify differences in the two key outcomes. Participants will complete baseline data collection (including medical history, medication use, and lower extremity venous assessment) before or shortly after radiofrequency ablation, undergo 30-day postoperative follow-up to evaluate bleeding events (such as minor bleeding or major bleeding requiring medical intervention), receive venous ultrasound at 3 months postoperatively to measure venous closure rate, and report any medication changes or adverse events during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, with a confirmed diagnosis of primary lower extremity varicose veins (CEAP classification C2-C6) based on clinical examination and duplex ultrasound.
* Underwent endovenous radiofrequency ablation (RFA) of the great saphenous vein as the primary intervention.
* Postoperatively, either: (a) continuously uses standard-dose oral antiplatelet drugs (e.g., aspirin 100mg/day, clopidogrel 75mg/day) or oral anticoagulant drugs (e.g., warfarin with INR maintained at 2.0-3.0, direct oral anticoagulants at standard therapeutic doses) as per clinical routine, or (b) does not use any antithrombotic drugs.
* Able to understand and comply with the follow-up schedule (including 30-day bleeding assessment and 6-month duplex ultrasound examination) and provide informed consent.

Exclusion Criteria:

* Presence of secondary varicose veins caused by deep vein thrombosis, venous malformation, or other vascular disorders.
* History of coagulation disorders (e.g., hemophilia, thrombocytopenia with platelet count <100×10⁹/L) or use of other antithrombotic agents (e.g., low-molecular-weight heparin, glycoprotein IIb/IIIa inhibitors) postoperatively.
* Major bleeding events (e.g., gastrointestinal bleeding, intracranial hemorrhage) within 3 months prior to RFA.
* Severe hepatic insufficiency (Child-Pugh class C), renal insufficiency (eGFR <30 mL/min/1.73m²), or other life-threatening systemic diseases.
* Unable to complete follow-up due to mental disorders, mobility limitations, or other reasons, or refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged ≥18 years with confirmed primary lower extremity varicose veins (CEAP classification C2-C6), validated by clinical examination and duplex ultrasound, who have undergone endovenous radiofrequency ablation (RFA) of the great saphenous vein as the primary treatment. Participants are stratified into three groups based on postoperative antithrombotic medication use per routine clinical practice: those taking standard-dose oral antiplatelet drugs, those using standard oral anticoagulants, and a control group without antithrombotic agents. Excluded individuals are patients with secondary varicose veins (e.g., due to deep vein thrombosis or venous malformations), coagulation disorders, postoperative non-oral antithrombotic use, major bleeding within 3 months before RFA, severe hepatic/renal insufficiency, life-threatening systemic diseases, or those unable to complete follow-up or provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
6-month postoperative venous closure rate | 6 month
6-month postoperative venous closure rate | 6-month

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] San Norberto Garcia EM, Merino B, Taylor JH, Vizcaino I, Vaquero C. Low-molecular-weight heparin for prevention of venous thromboembolism after varicose vein surgery in moderate-risk patients: a randomized, controlled trial. Ann Vasc Surg. 2013 Oct;27(7):940-6. doi: 10.1016/j.avsg.2013.03.006. PMID 23993109
- [Background] Gonzalez Ochoa AJ, Carrillo J, Manriquez D, Manrique F, Vazquez AN. Reducing hyperpigmentation after sclerotherapy: A randomized clinical trial. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):154-162. doi: 10.1016/j.jvsv.2020.06.019. Epub 2020 Jul 30. PMID 32739509
- [Background] Beyer-Westendorf J, Schellong SM, Gerlach H, Rabe E, Weitz JI, Jersemann K, Sahin K, Bauersachs R; SURPRISE investigators. Prevention of thromboembolic complications in patients with superficial-vein thrombosis given rivaroxaban or fondaparinux: the open-label, randomised, non-inferiority SURPRISE phase 3b trial. Lancet Haematol. 2017 Mar;4(3):e105-e113. doi: 10.1016/S2352-3026(17)30014-5. Epub 2017 Feb 16. PMID 28219692